CLINICAL TRIAL: NCT00813176
Title: One-Lung Ventilation in Morbidly Obese Patients:
Brief Title: One-Lung Ventilation in the Morbidly Obese Patient: Comparison of Double Lumen Versus Bronchial Blockers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier H Campos (Other)
Responsible Party: Sponsor-Investigator, Javier H Campos, Professor in Anesthesia, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200701755
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: Obesity; One-Lung Ventilation; Anesthesia; Thoracic; One-lung ventilation in the morbidly obese patient
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: prospective randomized study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double Lumen Endotracheal Tube (Active Comparator): We used a device called a double lumen tube ( DLT Broncho-Cath®). It is a bifurcated endotracheal tube designed to independently collapse the operated lung.
  Interventions: Device: Double Lumen Endotracheal Tube
- Arndt Bronchial Blocker (Active Comparator): We used a device called a bronchial blocker (9 Fr Arndt® blocker) along with a standard single-lumen tracheal tube (8.0-9.0 mm ID). The Arndt bronchial blocker is a single device, with a distal balloon that is passed thru the single lumen endotracheal once the patient is intubated. The Arndt bronchial blocker is designed to collapse the operated lung.
  Interventions: Device: Arndt Bronchial Blocker

INTERVENTIONS:
Device: Double Lumen Endotracheal Tube
  Arms: Double Lumen Endotracheal Tube
Device: Arndt Bronchial Blocker
  Arms: Arndt Bronchial Blocker

SUMMARY:
The purpose of this study is to determine whether the double-lumen endotracheal tube or the standard single-lumen tracheal tube, with an Arndt® blocker, is superior in providing one lung ventilation during thoracic surgery.

DETAILED DESCRIPTION:
The purpose of the study is to compare a double lumen tube versus the standard single-lumen tracheal tube, with an Arndt® blocker, in the morbidly obese patient who requires one-lung ventilation during surgery. The objects is to determine which device is best for intubation and is most effective in terms of optimal positioning of the device, of lung collapse, and quality of lung isolation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject undergoing thoracic or esophageal surgery requiring one-lung ventilation.
2. Subject is >18 years of age.
3. Subject's BMI > 35.

Exclusion Criteria:

1. Subject < 18 years of age.
2. Subject's BMI < 35.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier H Campos, MD, Principal Investigator — Iowa Health Care
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Double Lumen Endotracheal Tube: Double Lumen Endotracheal Tube This group was one arm of this research to determine the advantages of this group versus a comparative bronchial blocker group.
  We assessed 56 subjects and enrolled 50. A total of 6 were excluded because they did not meet criteria (4) or refused to participate (2).
- Arndt Bronchial Blocker: Arndt Bronchial Blocker We assessed 56 subjects and enrolled 50. A total of 6 were excluded because they did not meet criteria (4) or refused to participate (2).
Period: Overall Study
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Double Lumen Endotracheal Tube: Double Lumen Endotracheal Tube Device where lung collapse can be achieved by clamping one of the lumens (the operated lung) 25 subjects were enrolled in this group
- Arndt Bronchial Blocker: Arndt Bronchial Blocker in conjunction with a single lumen endotracheal tube. Device that allows collapse of one lung (the operated lung). 25 subjects were enrolled in this group
- Total: Total of all reporting groups
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Full Range); unit: years] | 52 [24 to 74] | 53 [23 to 85] | 52 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 11 | 12 | 23
double lumen tubes versus bronchial blockers [Count of Participants; unit: Participants] | 25 | 25 | 50
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index of obesity or being underweight. It is body weight divided by body height squared (BMI=kg/m^2)
  kg/m^2 | 39.9 (4.8) | 40.2 (4.5) | 40 (4.5)
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 114.5 (17.1) | 116.5 (22.4) | 115.6 (19.9)
Neck Circumference [Mean (Standard Deviation); unit: Centimeters] | 46 (4) | 47 (7) | 46.3 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Time Taken for Endotracheal Tube Placement Procedure.
Description: For each group, the time in minutes required for the anesthesiologist to successfully place the endotracheal tube.
  Intubation time was recorded as the time from when the tracheal tube passed the vocal cords until the anesthetist concluded that the DLT (Arm 1) or the single-lumen tube with the Arndt blocker (Arm 2) was correctly placed and optimal position was confirmed with the fiberoptic bronchoscope.
Time Frame: This measurement occurred after the patient was in the operating room and the randomization group was determined. This measurement began and ended during the intubation procedure.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Double Lumen Endotracheal Tube: Left-sided double lumen endotracheal tube Broncho-Cath®
- Arndt Bronchial Blocker: Arndt® blocker group: Intubation with a standard single-lumen tracheal tube (8.0-9.0 mm ID) followed by the passage of a 9 Fr Arndt® spherical blocker
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker
Number analyzed (Participants) | 25 | 25
minutes | 3.4 (1.8) | 4.1 (5.2)

2. Primary Outcome: Number of Participants in Which the Tube Was Successfully Positioned at First Attempt
Description: Number of participants in each group in which the tube was successfully positioned at first attempt
Time Frame: This data measure was occurred during surgery.
Measure: Count of Participants; unit: Participants
Groups:
- Double Lumen Endotracheal Tube: Double Lumen Endotracheal Tube
- Arndt Bronchial Blocker: Arndt Bronchial Blocker
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker
Number analyzed (Participants) | 25 | 25
Participants | 22 | 23

3. Secondary Outcome: Effectiveness of Lung Collapse
Description: For each group, the number of participants in which lung collapse was evaluated as: (i) good-complete collapse without surgical interference, (ii) fair-total collapse, but with residual air, and (iii) poor-no or partial collapse, lung inflated and interfering with the surgical exposure.
Time Frame: This measure occured during surgery just after intubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker
Number analyzed (Participants) | 25 | 25
Participants
  Good | 16 | 17
  Fair | 7 | 7
  Poor | 1 | 1
  Lung Colapse not Required | 1 | 0

4. Secondary Outcome: Time Required to Collapse the Lung
Description: For each group, the mean time for lung isolation/collapse was measured from the institution of one-lung ventilation to the time of total lung collapse.
Time Frame: This measurement occurred during surgery.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker
Number analyzed (Participants) | 25 | 25
Minutes | 18 (9.3) | 15.8 (9.6)

5. Secondary Outcome: Number of Participants With Successful Reinflation
Description: In each group, the number of Participants in which successful lung reinflation occurred.
Time Frame: This occurred during surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker
Number analyzed (Participants) | 25 | 25
Participants | 24 | 25

6. Secondary Outcome: Mean Intraoperative Oxygenation During One-lung Ventilation
Description: For each group, the mean intraoperative oxygenation (arterial partial pressure of oxygen measured by arterial blood gases) were taken during two-lung ventilation (baseline) and after 30 min of one-lung ventilation.
Time Frame: This measure occured during surgery.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker
Number analyzed (Participants) | 25 | 25
kPa | 16.8 (8.8) | 18.6 (10.3)

ADVERSE EVENTS:
Arm/Group | Double Lumen Endotracheal Tube | Arndt Bronchial Blocker
Serious Adverse Events (participants affected / at risk) | 3/25 | 2/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Lumen Endotracheal Tube (N=25) | Arndt Bronchial Blocker (N=25)
failure to intubate at first attempt (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) — failure to intubate at first attempt
(Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — there were no complications or adverse events related to this study
low PaO2 was seen in two patients one in each group and required Continuous positive airway pressure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — low Pao2 that was seen in one patient in each group and it was corrected with continuous positive airway pressure ventilation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes